CLINICAL TRIAL: NCT00594594
Title: A Multi-Centered, Randomized, Double-Blind, Placebo-Controlled Trial for Efficacy in the Use of Adjuntive Probiotic Therapy in Reducing Urinary Tract Infections in Those Individual With Spinal Cord Injury
Brief Title: Adjuntive Probiotic Therapy in Treating Urinary Tract Infections in Spinal Cord Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit enough patients to continue on with the study.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Dr. Gregor Reid, Lawson Health Research Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: R-06-213; HSREB 12845
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Spinal Cord Injury; Urinary Tract Infections
Keywords: spinal cord injury; urinary tract infection; probiotics; Lactobacilli
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Probiotic Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14
  Interventions: Other: Probiotic Lactobacillus GR-1 and RC-14

INTERVENTIONS:
Other: Probiotic Lactobacillus GR-1 and RC-14 — Two capsules of Lactobacillus GR-1 and RC-14 daily for 12 months

SUMMARY:
We hypothesize that probiotic Lactobacillus can augment antibiotic treatment of symptomatic urinary tract infection (UTI) in spinal cord injured patients, and also increase the time to the next episode of UTI.

DETAILED DESCRIPTION:
Subjects will be recruited from the outpatient population and 'alumni' of the Regional SCI Rehabilitation Programs in London (Parkwood Hospital/St Joseph's Health Care) and Hamilton (Hamilton Health Sciences Centre) Ontario.

Community living paraplegic and tetraplegic men and women (18 years and above) who present to their family physician or specialist with symptomatic UTI will be prescribed an antibiotic treatment for up to 14 days (using the drug of choice i.e. which the treating physician deems appropriate) and randomized to also receive by mouth two capsules containing placebo or probiotic Lactobacillus rhamnosus GR-1 and L. reuteri RC-14 daily.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* UTI
* > 18years
* Male and females
* Prescribed antibiotics

Exclusion Criteria:

* Patients who are participating in another clinical study involving pharmaceutical products.
* Patients who are participating in other urology clinical study.
* Patients taking yogurt containing probiotic lactobacilli during the period of the study.
* Females who are pregnant and/or planning to get pregnant during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Increase time to next UTI | 12 months

SECONDARY OUTCOMES:
Numbers of infections of any type occurring during probiotic treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Potter, MD FRCPC, Principal Investigator — St. Joseph's Health Care Centre, Parkwood Hospital, Lawson Health Research Institute; Gregor Reid, PhD, MBA, Study Director — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Keith Hayes, PhD, Study Chair — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Kingsley C Anukam, PhD, Principal Investigator — Lawson Health Research Institute, kanukam@uwo.ca
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Hayes KC, Bassett-Spiers K, Das R, Ethans KD, Kagan C, Kramer JL, Linsenmeyer T, Moore KN, Razvi H, Reid G, Walter JS, Wilson JW. Research priorities for urological care following spinal cord injury: recommendations of an expert panel. Can J Urol. 2007 Feb;14(1):3416-23. PMID 17324320